CLINICAL TRIAL: NCT03246061
Title: INTRACEPT: A Prospective, Randomized, Multi-Center Study of Intraosseous Basivertebral Nerve Ablation for the Treatment of Chronic Low Back Pain
Brief Title: INTRACEPT: Prospective, Randomized, Multi-center Study Intraosseous Basivertebral Nerve Ablation for Treatment of CLBP
Acronym: CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relievant Medsystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIP 0006
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: BVN Ablation vs Standard Care Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- BVN Ablation (Active Comparator): BVN ablation with continued standard care
  Interventions: Device: Intracept System
- Standard Care Control (Active Comparator): Continue with non-surgical standard care
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: Intracept System — BVN ablation using radiofrequency energy
  Arms: BVN Ablation
Other: Standard Care — Non-surgical standard care
  Arms: Standard Care Control

SUMMARY:
Prospective, open-label, 1:1 randomized controlled trial of Basivertebral nerve (BVN) Ablation arm vs Standard Care Control for the treatment of vertebrogenic chronic low back pain (CLBP). Participants in the the BVN Ablation arm will receive radiofrequency ablation of the BVN using the Intracept procedure for treatment of up to 4 vertebral bodies (L3 to S1). Participants in the Standard Care Control arm will continue on non-surgical standard care and will be offered optional crossover after 12 months of follow-up with follow-up of 6 months post crossover treatment.

The study had a pre-specified Interim Analysis with stopping rules for superiority when approximately 60% of the randomized participants have completed their 3-month primary endpoint study visit. An independent Data Safety Management Board (DSMB) reviewed the interim analysis results and recommended stopping enrollments for superiority and offering early crossover to the control arm participants.

DETAILED DESCRIPTION:
Participants in the BVN Ablation arm will be followed for 24 months following treatment. BVN Ablation arm participants will be approached to participate in a sub study of 3 additional years of follow-up at their 24 month visit (total of 5 years of follow-up).

Control arm subjects who were originally to be offered optional crossover treatment after the 12 month follow-up visit were offered crossover per the DSMB recommendation at a mean of 176.5 days.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature subjects at least 25 years of age
* Chronic lower back pain for at least 6 months
* Failure to respond to at least 6 months of non-operative conservative management

Exclusion Criteria:

* Radicular pain
* Current or history of spinal infection
* Modic changes at vertebral bodies other than L3 to S1
* Contraindication to MRI
* Pregnant, lactating or plan to become pregnant in next year
* Has life expectancy of less than 2 years
* Compensated injuries or ongoing litigation regarding back pain/injury, or financial incentive to remain impaired

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Garfin, MD, Principal Investigator — Independent
Locations (18):
- United States (18):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Barrow Brain and Spine, Phoenix, Arizona
  - Keck Medicine of USC, Los Angeles, California
  - Stanford Orthopaedic Surgery, Redwood City, California
  - Denver Back Specialists, Greenwood Village, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Drug Studies America, Marietta, Georgia
  - Beaumont Hospital, Royal Oak, Michigan
  - St Luke's Hospital, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Bassett Medical Center, Cooperstown, New York
  - University of Rochester, Rochester, New York
  - OrthoCarolina, Charlotte, North Carolina
  - Clinical Investigations, Edmond, Oklahoma
  - Pacific Sports and Spine, Eugene, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Precision Spine Center, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Trial results will be published at the completion of the trial
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: End of trial
Access Criteria: To be determined

REFERENCES:
- See also: INTRACEPT Study Website — http://intraceptstudy.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 420 patients screened for MRI Modic changes at levels L3 to S1 to achieve 140 enrollments. Patients with Modic changes at other levels or who had other primary etiologies for their low back pain (i.e. disc herniation, stenosis, facet joint) were excluded. An independent orthopedic surgeon medical reviewer confirmed eligibility prior to randomization. A pre-specified interim analysis was conducted when 60% of randomized patients completed their 3-month primary endpoint visit.
Groups:
- Basivertebral Nerve (BVN) Ablation: BVN ablation with non-surgical standard care
  Intracept System: BVN ablation
Period: Overall Study
Arm/Group | Basivertebral Nerve (BVN) Ablation | Standard Care Control
Started | 66 | 74
Interim Analysis | 51 | 53
Completed | 51 | 53
Not Completed | 15 | 21
Not completed — Still in follow-up | 15 | 21

BASELINE CHARACTERISTICS:
Groups:
- Basivertebral Nerve (BVN) Ablation: BVN ablation with standard care
  Intracept System: BVN ablation
- Standard Care Control: Continue standard care
- Total: Total of all reporting groups
Arm/Group | Basivertebral Nerve (BVN) Ablation | Standard Care Control | Total
Number analyzed (Participants) | 51 | 53 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (9.0) | 50.0 (11.1) | 50.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 26 | 25 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 49 | 48 | 97
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 53 | 104
Baseline Oswestry Disability Index (ODI) [Mean (Standard Deviation); unit: units on a scale] — Oswestry Disability Index (ODI) total score is on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The minimally clinically important difference for this tool is considered to be a 10 point reduction from baseline.
  units on a scale | 44.0 (11.8) | 48.1 (11.2) | 46.1 (11.3)
Baseline Visual Analogue Scale (VAS) [Mean (Standard Deviation); unit: units on a scale of 0 to 10] — Low Back Pain Visual Analog Scale (VAS). Participant indicated level of low back pain on a 10 point numeric scale with 0 being no pain and 10 being maximum pain. The published minimal clinically important difference for VAS is a 2 point reduction from baseline value.
  units on a scale of 0 to 10 | 6.51 (1.31) | 6.82 (1.34) | 6.67 (1.33)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Arms in Least Squared (LS) Mean Change in Oswestry Disability Index (ODI)
Description: Difference between arms in LS Mean change in ODI (baseline to 3 months post-treatment). ODI is measured on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The minimally clinically important difference for this tool is considered to be a 10 point reduction in ODI from a baseline in a patient.
  These data are for interim analysis of the primary endpoint. Data for later time points will be included in the current Outcome Measures as additional Rows, once available.
Time Frame: 3 months
Population: Interim Analysis N=104 (pre-specified interim analysis when approximately 60% of randomized participants complete their 3-month primary endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Basivertebral Never (BVN) Ablation: BVN ablation with standard care
  Intracept System: RF ablation
- Standard Care Control: Continue with standard care
Arm/Group | Basivertebral Never (BVN) Ablation | Standard Care Control
Number analyzed (Participants) | 51 | 53
units on a scale | -25.3 [-29.6 to -21.0] | -4.4 [-8.7 to -0.2]
Statistical Analysis 1: Comparison: Basivertebral Never (BVN) Ablation vs Standard Care Control; Estimates and p-value from an ANCOVA with a factor of treatment group and a covariate of baseline ODI score. Values have been adjusted for multiple imputation. Note: 3 month visit is computed as post-treatment for the RF Ablation Arm, and post-randomization for the Control Arm; Test type: Superiority; p < 0.001, ANCOVA — Interim Analysis p-value for significance of <0.025 for an overall alpha of 0.05

2. Secondary Outcome: Difference Between Arms in LS Mean Change in Visual Analog Scale (VAS)
Description: Difference between arms in LS Mean reduction in Visual Analog Scale (VAS) for low back pain from baseline to 3 months post treatment. VAS is a 10 point scale with 0 being no pain and 10 being worst imaginable pain. Participants are asked to indicate an x on the scale that corresponds to their perceived level of pain in their low back. The published minimal clinically important change in VAS is 2 points from baseline.
  These data are for interim analysis of the primary endpoint. Data for later time points will be included in the current Outcome Measures as additional Rows, once available.
Time Frame: 3 months post treatment / randomization
Population: Interim Analysis population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Basivertebral Nerve (BVN) Ablation | Standard Care Control
Number analyzed (Participants) | 51 | 53
units on a scale | -3.46 [-4.10 to -2.82] | -1.02 [-1.66 to -0.37]
Statistical Analysis 1: Comparison: Basivertebral Nerve (BVN) Ablation vs Standard Care Control; Test type: Superiority; p < 0.001, ANCOVA — Estimates and p-value from ANCOVA with a factor of treatment group and a covariate of baseline VAS score

ADVERSE EVENTS:
Time Frame: Enrollment through 24 month follow-up
Arm/Group | BVN Ablation | Standard Care Control
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/74
Other Adverse Events (participants affected / at risk) | 16/66 | 6/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BVN Ablation (N=66) | Standard Care Control (N=74)
Transient Leg Pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (2) — Temporary leg pain resolved in mean of 42 days
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) — Post anesthesia related urinary retention. Resolved with catheterization.
Incisional Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Post procedure incision region discomfort
Ongoing low back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Disc Herniation (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Incomplete Procedure (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Inability to access

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT03246061/Prot_SAP_000.pdf